CLINICAL TRIAL: NCT07014800
Title: Multi-frequency MR Elastography Based Tomoelastography: Additional New Imaging Tool for Postoperative Pancreatic Fistula Risk Stratification
Brief Title: Tomoelastography in Predicting Postoperative Pancreatic Fistula
Acronym: POPF
Status: Completed | Type: Observational
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Siya Shi, clinical doctor, First Affiliated Hospital, Sun Yat-Sen University
Other Study IDs: FirstSunYetSen123
Record Dates: First submitted 2025-06-03; First posted 2025-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Pancreatectomy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- patients with postoperative pancreatic fistula
- patients without postoperative pancreatic fistula

SUMMARY:
Postoperative pancreatic fistula (POPF) is a prevalent and severe complication of pancreaticoenteric anastomosis; however, its accurate preoperative prediction is challenging. Multi-frequency MR elastography-based tomoelastography can quantify pancreatic mechanical properties (stiffness and fluidity), thus further improving the predictive performance of conventional MRI for postoperative pancreatic fistulas.

ELIGIBILITY:
Inclusion Criteria: Participants diagnosed with postoperative pancreatic fistula who underwent both preoperative multi-frequency MRE and pancreaticoenteric anastomosis were included in the study.

-

Exclusion Criteria:

without appropriate image quality； without available pathological data

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Participants who underwent both preoperative multi-frequency MRE and pancreaticoenteric anastomosis were included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 157 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-07-31 (Actual); Study Completion 2024-07-31 (Actual)

PRIMARY OUTCOMES:
Postoperative pancreatic fistula | The participants were routinely examined on days 1, 3, 5, and 7 after surgery to determine fluid volumes and serum amylase levels.
  Any measurable drainage of amylase levels above three times the upper limit of the normal amylase level on or after the third postoperative day was considered the essential threshold of diagnosing postoperative pancreatic fistula.

CONTACTS AND LOCATIONS:
Locations (1):
- Shi Siya, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No
All data generated for this study are from the corresponding author upon reasonable request.